CLINICAL TRIAL: NCT02381119
Title: The Personalized Dietary Advice Services: Effects of Use by the Dietician on Health Status of Diabetes Type 2 Patients
Brief Title: Effects of Personalized Dietary Advice on Health Status of Diabetes Type 2 Patients
Acronym: PDA(4)T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Vitas (Unknown); SwissAnalysis (Unknown)
Responsible Party: Principal Investigator, W.J. Pasman, Project leader Clinical studies, TNO
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P9618
Record Dates: First submitted 2015-02-24; First posted 2015-03-06 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: dietary services; personalized advice; biological markers
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Algorithms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized advice (Experimental): Dietitian provides Personalized dietary advice (based on genetic, blood and food intake profiles) (the type of advice is the intervention)
  Interventions: Behavioral: Personalized Dietary Advice Services
- Regular care (Active Comparator): Dietitian provides regular care for diabetes type 2 (regular advice is the control condition)
  Interventions: Behavioral: Regular care

INTERVENTIONS:
Behavioral: Personalized Dietary Advice Services — This Personalized Dietary Advice is based on markers for nutrition status and SNPs (single nucleotide polymorphisms).
  This advice is given via Personalized Dietary Advice Services, in which health data of the client can be entered and will be translated into advice on intake of specific nutrients or food categories.
  Other Names: Algorithms for personalized dietary advice; Food4Me algorithms; Dietary advice based on individual health status
  Arms: Personalized advice
Behavioral: Regular care — The control group will receive usual advice for diabetes type 2 from the dietician. However, after the end of the study participants in the control group will be offered the opportunity to receive the Personalized Dietary Advice from their dietician, as based on the parameters measured during the study.
  Arms: Regular care

SUMMARY:
This study addresses the challenge of increasing compliance with dietary recommendations and guidelines among diabetes type 2 patients by introducing professional dietary advice based on individual requirements.

The objective of this study is to assess the effect of the Personalized Dietary Advice Services (PDAS) after a three month intervention on established markers of nutritional and health status in diabetes type 2 patients (HbA1c, glucose, insulin). Besides, the effect of the PDAS on perceived health status of diabetes type 2 patients will be assessed.

DETAILED DESCRIPTION:
This study will be a randomized control trial studying the effect of personalized dietary advice services on established markers of nutrition and health status of diabetes type 2 patients. This dietary advice will be based on individual genetic, blood and food intake profiles, which will be measured at the start of the study.

The dietitian will provide this personalized dietary advice, during the regular patient visits. In the control group, the dietitian will give the regular dietary advice.

The study will start with a run-in period of two weeks, during which baseline measures will be done. After the run-in period, the three-month study will start with a first dietary consult during which the dietitian will use the personalized dietary advice services for providing dietary advice in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80 years;
* Stable BMI 25-35 kg/m2
* Diabetes type 2 as diagnosed by the General Practitioner (GP), based upon:
* Fasting glucose > 6.9 mmol/l on two different days or one measurement of non-fasting glucose > 11.0 mmol/l in combination with symptoms of hyperglycemia
* Healthy as assessed by the health and lifestyle questionnaire (P9607 F02; in Dutch);
* Voluntary participation;
* Informed consent signed;
* Willing to comply with the study procedures;
* Willingness to share pseudonymized data on food intake with external party MijnEetmeter (food intake app provider)
* Willingness to share pseudonymized data on physical activity with external party Medisana (provider of activity tracker)
* Willingness to share pseudonymized data on food intake, blood glucose, blood cholesterol, blood pressure, physical activity and body weight with the Nutrition Research Cohort (NRC) database
* Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for 15 years.
* Have a desktop or laptop with internet access at home.

Exclusion Criteria:

* Use of concomitant medication including medication known for its effects the main study parameters, except for medication for diabetes type 2, cholesterol or blood pressure;
* Use of insulin or Sulfonyl Urea derivatives;
* Slow onset type 1 diabetes;
* Diabetes occurring after several attacks of pancreatitis known as pancreatic diabetes;
* (Having a history of a) medical condition that might significantly affect the study outcome as judged by the medical investigator and health and life style questionnaire. This includes diabetes type 1, gastrointestinal dysfunction, diseases related to inflammation or allergy, or a psychiatric disorder;
* Following a medically prescribed diet, other than dietary advice for diabetes type 2;
* Use of nutritional supplements that could influence the study outcome, including vitamin supplements, fish oil and/or omega fatty acids;
* Physical, mental or practical limitations in using computers;
* Alcohol consumption > 21 (women) - 28 (men) units/week;
* Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre-study screening;
* Recent blood donation (< 1 month prior to the start of the study);
* Not willing to give up blood donation during the study;
* Not having a general practitioner;
* Personnel of TNO in Zeist and Soesterberg and their partners.
* Not willing to accept information-transfer concerning study participation, or health-related information, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from the participant's general practitioner.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
change in fasting plasma glucose | week -2 (run-in period) and week 13 (end of study)
  blood glucose levels after an overnight fast (not eating or drinking for at least 8 hours)
change in HbA1c levels | week -2 (run-in period) and week 13 (end of study)
  representing change in long-term blood glucose levels
change in fasting insulin levels | week -2 (run-in period) and week 13 (end of study)
  blood insulin levels after an overnight fast (not eating or drinking for at least 8 hours)

SECONDARY OUTCOMES:
change in body weight | week -2 (run-in period), week 0, week 4, week 8 and week 13 (end of study)
  also used for calculation of body mass index (BMI)
change in waist-to-hip ratio | week -2 (run-in period), week 0, week 4, week 8 and week 13 (end of study)
  ratio between waist and hip circumference as measured by the dietitian
change in blood pressure | week -2 (run-in period), week 0, week 4, week 8 and week 13 (end of study)
  as measured by the dietitian
change in subjective quality of life as assessed with RAND-36 questionnaire | week 0 (baseline) and week 13 (end of study)
change in vitality as assessed with a vitality questionnaire (Vita-16) | week 0 (baseline) and week 13 (end of study)
change in physical activity as assessed with a physical activity questionnaire | week 0 (baseline) and week 13 (end of study)
user experiences with personalized dietary advice services as assessed with a questionnaire | week 13 (end of study)
change in blood cholesterol levels | week 0 (baseline), week 4, week 8 and week 13 (end of study)
  change in total cholesterol as well as HDL, LDL and triglyceride levels
change in biomarkers for food intake | week -2 (run-in period) and week 13 (end of study)
  change in blood levels representing food intake
change in levels of non-esterified fatty acids in blood | week -2 (run-in period) and week 13 (end of study)
20 nutrition-related SNPs (single nucleotide polymorphisms) | week -2 (run-in period)
  Genetic state

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (8):
  - Diëtistenpraktijk Sylvia van Daalen, Arnhem, Gelderland
  - Diëtistenpraktijk Verhoeven & Bac, Barendrecht, South Holland
  - independent practice Willy Gilbert, Dordrecht, South Holland
  - Diëtistenpraktijk Jansen-Sloot, Gorinchem, South Holland
  - Diëtistenpraktijk Care & Cure, Hillegom, South Holland
  - Diëtistenpraktijk MirjaM - Leefstijl & Dieet, Sassenheim, South Holland
  - Diëtistenpraktijk Dieetistopsport, Zoetermeer, South Holland
  - Netherlands Organisation for Applied Scientific Research (TNO), Zeist, Utrecht